CLINICAL TRIAL: NCT07244874
Title: A Single Arm, Phase II Study of Sacituzumab Tirumotecan（Sac-TMT） Combined With Toripalimab for First-line Treatment of PD-L1 Positive Unresectable Locally Advanced/Metastatic Triple Negative Breast Cancer (a/mTNBC)
Brief Title: Sac-TMT Combined With Toripalimab for First-line Treatment of PD-L1 Positive a/mTNBC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Southwest Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SKB264-IIT-004
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-07

CONDITIONS: TNBC - Triple-Negative Breast Cancer; PD-L1 Positive
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sacituzumab Tirumotecan + Toripalimab (Experimental)
  Interventions: Drug: Sacituzumab tirumotecan; Drug: Toripalimab

INTERVENTIONS:
Drug: Sacituzumab tirumotecan — 5mg/kg, Q2W
Drug: Toripalimab — 240mg，Q3W

SUMMARY:
This study is aimed to evaluate the efficacy and safety of Sacituzumab Tirumotecan combined with Toripalimab for first-line treatment of PD-L1 positive unresectable Locally Advanced/metastatic triple negative breast cancer (a/mTNBC).

ELIGIBILITY:
Inclusion Criteria:

1. Female patients with breast cancer aged >= 18 years.
2. Based on the pathological report of the latest biopsy or other pathological specimens, the histology and/or cytology are confirmed as invasive breast cancer, and the following conditions are met: a) Pathological classification: ER <= 10%, PR <= 10%; HER2 negative (IHC 0, 1+, 2+and FISH negative); Note: Subjects with initial histopathological diagnosis of HR>10% or HER2+breast cancer and recent pathological findings of metastatic lesions meeting the above conditions are allowed to be included in the study. b) Tumor staging: locally advanced, recurrent, or metastatic tumors that cannot be surgically removed; Note: Patients who have received perioperative treatment in the past are required to have a disease-free survival period of >= 6 months;
3. ECOG overall state is 0-1.
4. Have not received systematic treatment for advanced diseases.
5. There are tissue samples available for PD-L1 testing, and the test results show PD-L1 positive: CPS >= 1.
6. The expected survival period is not less than 3 months.
7. According to the RECIST v1.1 standard, there must be at least one measurable lesion present.
8. Having sufficient organ and bone marrow function (without receiving blood transfusion, recombinant human thrombopoietin or colony-stimulating factor therapy within 2 weeks prior to the first administration), defined as follows: a) Blood routine: neutrophil count (NEUT #) >= 1.5 × 10^9/L; platelet count (PLT) >= 100 × 10^9/L; hemoglobin >= 90g/dL; b) Liver function: Aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP) <= 2.5 x upper limit of normal (ULN); Total bilirubin (TBIL) <= 1.5 × ULN; For patients with liver metastases, ALT and AST should be <= 5 × ULN, and TBIL should be <= 2 × ULN; For patients with liver or bone metastases, ALP <= 5 × ULN; c) Renal function: creatinine clearance rate (Ccr) >= 60ml/min; d) Coagulation function: International normalized ratio (INR), activated partial thromboplastin time (APTT), and prothrombin time (PT) <= 1.5 × ULN; e) Cardiac function: Echocardiography (ECHO) or multi circuit controlled acquisition (MUGA) scan shows left ventricular ejection fraction (LVEF) >= 50%;
9. Patients must recover from all toxicity caused by previous treatment (to <= grade 1, evaluated based on CTCAE 5.0, or meet the inclusion criteria of the protocol), except for hair loss and vitiligo.
10. Patients with negative serum pregnancy test results and those with fertility potential must agree to use effective non hormonal contraceptive methods during treatment and for at least 6 months after the last use of the test drug.
11. Voluntarily joining this study, signing informed consent, having good compliance, and willing to cooperate with follow-up.

Exclusion Criteria:

1. Patients with central nervous system metastases.
2. Received radiotherapy, endocrine therapy, chemotherapy, surgical treatment (excluding local puncture or biopsy) or molecular targeted therapy during the recurrence/metastasis stage.
3. Participated in clinical trials of other drugs within 4 weeks prior to enrollment.
4. Previously treated with anti-PD-1, anti-PD-L1, anti-PD-L-2, or anti-CTLA-4 antibodies, or any other antibodies or drugs that specifically target T cell co stimulatory or checkpoint pathways.
5. Previously used treatment targeting TROP2 and/or topoisomerase I inhibitors.
6. Other malignant tumors within the past 5 years, excluding cured cervical carcinoma in situ, basal cutaneous carcinoma, or squamous cell carcinoma of the skin.
7. Known history of allergies to the drugs and their components in this protocol.
8. Human immunodeficiency virus (HIV) test is positive or there is a history of acquired immunodeficiency syndrome (AIDS); Known active syphilis infection.
9. History of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
10. Vaccination with live vaccine within 30 days prior to the first study administration.
11. History of (non infectious) interstitial lung disease (ILD) or non infectious pneumonia requiring steroid treatment, current ILD or non infectious pneumonia, or suspected ILD or non infectious pneumonia that cannot be excluded by imaging examination during screening; Clinical severe lung damage caused by concurrent lung diseases, including but not limited to any underlying lung disease (such as pulmonary embolism, severe asthma, severe chronic obstructive pulmonary disease, restrictive lung disease, pleural effusion, etc. within 3 months prior to administration) or any autoimmune, connective tissue, or inflammatory disease that may affect the lungs (i.e. rheumatoid arthritis, Sjogren's syndrome, sarcoidosis, etc.), or previous total pneumonectomy.
12. Patients with active autoimmune diseases that need systematic treatment in the past two years (hormone replacement therapy is not considered as systematic treatment, such as type I diabetes, hypothyroidism requiring only thyroid hormone replacement therapy, adrenal or pituitary insufficiency requiring only physiological dose of glucocorticoid hormone replacement therapy).
13. Active infections requiring systemic treatment within 2 weeks prior to the first administration.
14. ccording to the investigator's judgment, there are concomitant diseases that seriously endanger the patient's safety or affect the patient's completion of the study, including but not limited to high blood pressure beyond the control of drugs, serious diabetes, active infection, etc.
15. There is a recorded history of severe dry eye syndrome, severe meibomian gland disease and/or blepharitis, or corneal diseases that hinder delayed corneal healing.
16. Pregnant and lactating female patients, female patients with fertility and positive baseline pregnancy test results, and female patients of childbearing age who are unwilling to take effective contraceptive measures during the trial drug treatment period and the last 6 months of medication..
17. The researchers believe that the patient is not suitable to participate in any other circumstances of this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Enrollment: 41 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-01-30 (Estimated); Study Completion 2029-07-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to approximately 15 months

SECONDARY OUTCOMES:
Progression-Free-Survival | Up to approximately 15 moths
Duration of Response | Up to approximately 15 months
Overall Survival | Up to approximately 4 years
adverse events | Up to approximately 15 months

IPD SHARING:
Plan to Share IPD: No